CLINICAL TRIAL: NCT03647371
Title: Thyromental Height Test as a New Method for Prediction of Difficult Intubation Using Videolaryngoscopy
Brief Title: TMHT - Difficult Intubation Prediction Using Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TMHT-03
Record Dates: First submitted 2018-08-05; First posted 2018-08-27 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Predictive Value of Tests; Intubation
Keywords: Difficult Intubation; Thyromental Height Test; Videolaryngoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macintosh laryngoscope (Other): direct laryngoscope - laryngoscope with Macintosh blade
  Interventions: Procedure: Macintosh laryngoscopy
- McGrath videolaryngoscope (Other): McGrath Videolaryngoscope
  Interventions: Procedure: McGrath MAC video laryngoscopy

INTERVENTIONS:
Procedure: Macintosh laryngoscopy — intubation with MAcintosh laryngoscopy after anesthetic induction
  Arms: Macintosh laryngoscope
Procedure: McGrath MAC video laryngoscopy — intubation with McGrath MAC videolaryngoscopy after anesthetic induction
  Arms: McGrath videolaryngoscope

SUMMARY:
The purpose of this study is to assess the usefulness of the Thyromental Height Test in prediction of difficult intubation using videolaryngoscopy and double lumen endotracheal tubes in patients scheduled for elective thoracic procedures.

DETAILED DESCRIPTION:
Successful and fast intubation are crucial for the safety of general anaesthesia. Failed intubation and acute hypoxia remain among the major contributing factors of anaesthesia related deaths. Difficult intubation prevalence in literature is very inconsistent and varies between 1.5-20% of cases in general population, to even 50% in obese Thai population.

There is a number of anthropometric scales and tests used for predicting difficult intubation. However, none of them appears to be sensitive and specific enough to effectively predict difficult intubation.

Recently, simple and non-invasive test predicting difficult intubation was introduced-thyromental height test (TMHT). It shows promise as a more effective substitution for frequently cited anthropometric measures. It is based on the height between the anterior border of the thyroid cartilage and the anterior border of the mentum, measured while the patient lies in the supine position with closed mouth The main objective of the trial is to assess the clinical usefulness of TMHT in prediction of difficult intubation using videolaryngoscopy and double lumen endotracheal tubes in patients scheduled for elective thoracic surgical procedures. The secondary aim is to evaluate usefulness of other commonly used predictive tests associated with difficult intubation.

During routine, preoperative anaesthetic visit thyromental height, thyromental distance, sternomental distance and Mallampati scale score are assessed. Then, during videolaryngoscopy and intubation, score in Cormack-Lehane scale and occurrence of difficult intubation are noted.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective thoracic procedures, requiring general anaesthesia, videolaryngoscopy and intubation with a Robert-Shaw type double lumen endotracheal tubes
* written, informed consent for participation in the trail
* older than 18 years

Exclusion Criteria:

* emergency procedures
* visible anatomic abnormalities
* patients scheduled for awake fibre optic intubation
* lack of consent for participation in the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Thyromental height | From August 6 2018 to August 5 2019.
  The height between the anterior border of the thyroid cartilage (on the thyroid notch just between the 2 thyroid laminae) and the anterior border of the mentum (on the mental protuberance of the mandible), in supine position with mouth closed, measured with a depth gauge during routine preoperative anaesthetic visit.

SECONDARY OUTCOMES:
score in Cormack-Lehane scale | From August 6 2018 to August 5 2019.
  During videolaryngoscopy the laryngeal view is graded in Cormack-Lehane Scale by the laryngoscopist. Grade I is assigned when the glottis is fully visible, grade II when the glottis is partially visible, grade III when only the epiglottis is visible and grade IV when neither glottis nor epiglottis is visible.
Thyromental distance | From August 6 2018 to August 5 2019.
  The distance between the thyroid prominence and the most anterior part of the mental prominence of the mandible, measured with a standard centigrade ruler as the distance in centimetres with the patient in supine position, head fully extended, mouth closed, during routine preoperative anaesthetic visit.
Sternomental distance | From August 6 2018 to August 5 2019.
  The distance in centimetres between the superior border of the manubrium sterni and the bony point of the mentum, with the patient in supine position, head fully extended, mouth closed, measured with a standard centigrade ruler, during routine preoperative anaesthetic visit.
core in modified Mallampati test | From August 6 2018 to August 5 2019.
  The oropharyngeal view is assessed in sitting position, mouth maximally opened, tongue protruded, without phonation, measured during routine preoperative anaesthetic visit.
distance of mouth opening | From August 6 2018 to August 5 2019.
  Measured as a distance between the lower and upper incisors with a tape measure (Standard, Hoechstmas, Sulzbach, Germany) as a distance in centimetres. Patients are in sitting position with mouth maximally opened, tongue retracted and without phonation.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiołek, MD PhD, Study Director — Medical University of Silesia; Szymon Białka, MD, Study Chair — Medical University of Silesia
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No